CLINICAL TRIAL: NCT04620473
Title: Anlotinib Hydrochloride Combined With Capeox in the Neoadjuvant Treatment of Locally Advanced Rectal cancer-a Prospective, Open, Single Center and Randomized Controlled Phase Ⅱ Clinical Trial
Brief Title: Anlotinib Hydrochloride Combined With Capeox in the Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No approval from ethical committee
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Principal Investigator, Cai Zhenghao, Attending surgeon of gastrointestinal surgery, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai Minimally Invasive Surgery Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISC-Anlotinib+Capeox
Record Dates: First submitted 2020-10-29; First posted 2020-11-09 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Neoadjuvant Treatment; Rectal Cancer; Anlotinib
Keywords: Neoadjuvant Treatment; Rectal cancer; Anlotinib
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anlotinib+Capeox (Experimental): neoadjuvant treatment with Anlotinib hydrochloride combined with Capeox
  Interventions: Drug: Anlotinib+Capeox
- Capeox (Active Comparator): neoadjuvant treatment with Capeox
  Interventions: Drug: Capeox

INTERVENTIONS:
Drug: Anlotinib+Capeox — to use Anlotinib hydrochloride combined with Capeox in the neoadjuvant treatment of locally advanced rectal cancer
  Arms: Anlotinib+Capeox
Drug: Capeox — to use Capeox in the neoadjuvant treatment of locally advanced rectal cancer
  Arms: Capeox

SUMMARY:
Prospectively Investigate the effectiveness and safety of anlotinib hydrochloride combined with Capeox in neoadjuvant treatment of patients with locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily join the study and sign an informed consent form, have good compliance and cooperate with follow-up;
2. Male or female patients between the ages of 18-75;
3. Patients diagnosed as rectal adenocarcinoma by histology or cytology;
4. Stage: Locally advanced stage (T3-4N0M0 or T1-4N+M0);
5. Evaluation of middle and low rectal cancer with the lower pole of the tumor less than 12 cm from the anal margin by MRI;
6. Have not received other anti-angiogenic drugs or chemotherapy drugs in the past;
7. ECOG (Eastern US Cooperative Oncology Group) score: 0-1 points;
8. Has sufficient organ and bone marrow function

Exclusion Criteria:

1. Other malignant tumors that have appeared or are currently suffering from within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) ) And T1 (tumor infiltration basement membrane)];
2. A distant transfer occurs;
3. Those who have multiple factors that affect oral medications (such as inability to swallow, chronic diarrhea, etc.);
4. Accompanied by pleural effusion or ascites, causing respiratory syndrome (NCI-CTC AE V5.0 grade ≥ 2 dyspnea);
5. Patients with any severe and/or uncontrollable disease；
6. Patients with gastrointestinal diseases with bleeding tendency (such as active gastrointestinal ulcers) or patients determined by the researcher to cause gastrointestinal bleeding, perforation or obstruction
7. Patients whose imaging shows that the tumor has invaded the tissues around important blood vessels or the investigator judges that the tumor is likely to invade important blood vessels and cause fatal bleeding during the follow-up study;
8. Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before grouping;
9. Regardless of the severity, patients with any signs of bleeding or medical history; within 4 weeks before grouping, patients with any bleeding or bleeding events NCI-CTC AE V5.0 grade ≥ 3, unhealed wounds, ulcers Or fracture
10. Those who have had arterial/venous thrombotic events within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism;
11. People with a history of psychotropic drug abuse and unable to quit or have mental disorders;
12. Participated in other anti-tumor drug clinical trials within four weeks;
13. According to the judgment of the investigator, those with concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study;
14. Female patients who are pregnant or breastfeeding;
15. Known hypersensitivity to any study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | an average of three months
  Refers to the proportion of subjects whose tumors have shrunk to a certain amount and maintained for a certain period of time in the FAS concentration, including CR and PR cases

SECONDARY OUTCOMES:
Pathological complete response rate | one month after surgery
  Refers to the pathological examination of primary tumors and lymph node surgical specimens without residual infiltrating tumor cells (ypT0N0)
R0 resection rate | one month after surgery
  Refers to the surgically removed tissue without residual cancer cells
Local disease recurrence time | 3 years after surgery
  Refers to the tumor reappearing at or near the same site as the primary cancer. The starting time is the first day after surgery.
Overall survive | 3 years after surgery
  Refers to the time from the start of randomization to death due to any cause. The starting time is the first day after surgery.
Disease-free survival rate | 3 years after surgery
  It refers to the time from the beginning of randomization to the incurable resection, local recurrence or metastasis, or death from any cause. The starting time is the first day after surgery.
Postoperative complications | one month after surgery
  Postoperative complications

IPD SHARING:
Plan to Share IPD: Undecided